CLINICAL TRIAL: NCT07225322
Title: Low Intensity Focused Ultrasound in Autism Spectrum Disorder
Brief Title: Low Intensity Focused Ultrasound in ASD
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); COBRE in Neurodevelopment and its Disorders (CNDD) (Unknown)
Responsible Party: Principal Investigator, Kevin Caulfield, Assistant Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00146822; 5P20GM148302 (NIH)
Record Dates: First submitted 2025-09-04; First posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Active LIFU (Experimental)
  Interventions: Device: Active LIFU

INTERVENTIONS:
Device: Active LIFU — In this open label study, all participants will receive active LIFU

SUMMARY:
This study investigates the safety and potential efficacy of personalized, image-guided low intensity focused ultrasound (LIFU) targeting the thalamus in individuals with Autism Spectrum Disorder (ASD). The study evaluates behavioral, neuroimaging, and electrophysiological outcomes following LIFU stimulation using a non-invasive device.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-25
* Diagnosis of ASD (DSM-5)
* Full Scale IQ > 70
* Verbal communication
* Stable medication for ≥1 month
* Ability to consent or assent with guardian consent

Exclusion Criteria:

* MRI or LIFU contraindications
* Recent investigational drug/device use
* Neurological illness (e.g., epilepsy, TBI)
* Substance use disorder
* Sensory/motor impairments preventing task completion

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Social Responsiveness Scale, Second Edition (SRS-2) | Baseline (Visit 1) to post-stimulation (Visit 7, within 1 week of last stimulation; Visit 8, within 1 month of last stimulation)

SECONDARY OUTCOMES:
Penn Emotion Identification Task | Baseline (Visit 1) to post-stimulation (Visit 7, within 1 week of last stimulation; Visit 8, within 1 month of last stimulation)
Electroencephalography (EEG) in the alpha (8-12Hz) frequency band | Baseline (Visit 1) to post-stimulation (Visit 7, within 1 week of last stimulation)
Radiological MRI Safety Scans (T1, T2, diffusion scans, read for abnormalities) | Baseline (Visit 1) to post-stimulation (Visit 7, within 1 week of last stimulation)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Caulfield, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- MUSC Brain Stimulation Offices, Charleston, South Carolina, United States